CLINICAL TRIAL: NCT00004095
Title: Phase I Trial of Irinotecan (CPT-11) and Gemcitabine in Patients With Solid Tumors
Brief Title: Irinotecan Plus Gemcitabine in Treating Patients With Unresectable or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 98X3; NU-98X3; P-UPJOHN-976475157; NCI-G99-1588
Record Dates: First submitted 1999-12-10; First posted 2003-05-07 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Bladder Cancer; Breast Cancer; Colorectal Cancer; Kidney Cancer; Lung Cancer; Pancreatic Cancer
Keywords: stage IV colon cancer; stage IV breast cancer; recurrent breast cancer; recurrent non-small cell lung cancer; recurrent pancreatic cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; stage IV renal cell cancer; recurrent renal cell cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer; recurrent bladder cancer; stage IV bladder cancer; stage IV non-small cell lung cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Kidney Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Carcinoma, Non-Small-Cell Lung; Rectal Neoplasms; Carcinoma, Renal Cell; Small Cell Lung Carcinoma | interventions — Gemcitabine; Irinotecan

ARMS (1):
- Irinotecan Plus Gemcitabine (Experimental)
  Interventions: Drug: gemcitabine hydrochloride; Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining irinotecan and gemcitabine in treating patients who have unresectable or metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose (MTD) and the principal toxicities of irinotecan and gemcitabine in patients with surgically unresectable or metastatic solid tumors.
* Determine if the principal toxicities and MTD of this combination regimen are affected by drug sequencing in this patient population.
* Determine the potential for gemcitabine to alter the pharmacokinetic characteristics when administered with irinotecan in these patients.
* Describe the influence effected by varying the administration sequence of this combination regimen in this patient population.
* Obtain preliminary data regarding efficacy of this combination regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive irinotecan IV over 90 minutes followed by gemcitabine IV over 30 minutes on days 1 and 15. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity. Once the maximum tolerated dose (MTD) is reached, patients receive subsequent doses of the inverse sequence of the combination drugs until a new MTD is determined.

Cohorts of 3-6 patients receive escalating doses of irinotecan and gemcitabine until the MTD is reached. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicities.

Patients are followed every 3 months until death.

PROJECTED ACCRUAL: At least 12 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic or surgically unresectable solid tumor, having received the following maximum number of prior therapies for advanced disease:

  * Bladder cancer - no more than 1 prior therapy
  * Breast cancer - no more than 2 prior therapies
  * Colorectal cancer - no more than 1 prior therapy
  * Kidney cancer - no prior therapy
  * Lung cancer - no more than 1 prior therapy
  * Pancreatic cancer - no prior therapy
* Bidimensionally measurable disease outside a previously irradiated field

  * At least 2 cm x 2 cm
* No known bone metastases
* CNS involvement allowed if successfully controlled by surgery or radiotherapy and not requiring corticosteroids
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Menopausal status:

* Not specified

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL regardless of liver involvement secondary to tumor
* SGOT no greater than 3 times upper limit of normal (ULN) (no greater than 5 times ULN if liver metastases present)
* No known Gilbert's disease

Renal:

* Creatinine no greater than 1.8 mg/dL
* Calcium less than 12.0 mg/dL

Cardiovascular:

* No myocardial infarction within the past 6 months
* No congestive heart failure requiring therapy

Other:

* No active uncontrolled bacterial, viral (including HIV), or invasive fungal infection
* No psychiatric disorders that would prevent compliance
* No other malignancy within the past 5 years except adequately treated basal or squamous cell skin cancer or carcinoma in situ of the cervix
* No history of seizures
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent sargramostim (GM-CSF)
* No concurrent immunotherapy

Chemotherapy:

* No prior irinotecan, topotecan, or gemcitabine
* Prior adjuvant chemotherapy allowed, if at least 1 year between last dose of adjuvant chemotherapy and recurrence of cancer
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy to less than 30% of bone marrow
* No prior whole pelvic radiotherapy
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics

Other:

* No concurrent phenytoin, phenobarbital, or other antiepileptic prophylaxis

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 1999-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Al B. Benson, MD, FACP, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Result] Wisinski KB, Mulcahy MF, Newman S, et al.: A phase I study of irinotecan and gemcitabine in solid tumors. [Abstract] American Society of Clinical Oncology 2007 Gastrointestinal Cancers Symposium, 19 -21 January 2007, Orlando, Florida A-140, 2007.